### Nurses Stress Self-Care Educational Program (NSSCEP)

**Teaching Quid** 

22/8/2025

### NURSES' STRESS SELF CARE EDUCATIONAL PROGRAM

### DAY ONE / 2 HOURS

| Session 1: Self-Care for Nurses: Managing Occupational Stress and Preventing Burnout | | | |
|---|---|---|---|
| Objective | Content (Topics) | Materials/Aids | Teaching strategy |
| Define burnout and stress, list three sources, explain two effects on performance. | <ol> <li>Welcome note and program overview.</li> <li>Introduction to occupational stress and burnout</li> <li>Workshop Objectives</li> <li>Key Definitions of Occupational Stress and Burnout</li> <li>Effects of Stress on the Body and Mind</li> <li>The Importance of Self Stress Management Programme</li> </ol> | Laptop, digital projector, flip charts, reflection journal. | |
| Session2: Strengthening | Your Inner Resources: A Resili | ence and Copin | g Workshop |
| Objective | Content (Topics) | Materials/Aids | Teaching strategy |
| support to reduce burnout through improved communication and trust among colleagues, which has been shown to enhance nurse well-being | <ol> <li>Stress Management Techniques <ul> <li>Deep breathing exercises</li> <li>Progressive muscle relaxation</li> <li>Time management skills</li> <li>Grounding techniques</li> </ul> </li> <li>Resilience Training <ul> <li>Developing an optimistic outlook</li> <li>Problem-solving skills</li> <li>Building a support network</li> <li>Finding Meaning and Purpose:</li> </ul> </li> <li>Self-Compassion Practices</li> <li>Cognitive Restructuring</li> </ol> | Flip charts, communication skill checklist, reflection worksheets. | Interactive lecture, paired listening practice, empathy role-play, group discussion, mentorship planning. |

### NURSES' STRESS SELF CARE EDUCATIONAL PROGRAM

### DAY TOW / 2 HOURS

| Session 3: Reframing Stressful Thoughts with Positive Thinking | | | |
|---|---|---|---|
| Objective | Content (Topics) | Materials/Aids | Teaching strategy |
| Improve psychological | 1. Develop an attitude of | Flip charts, | Thought reframing |
| resilience by recognizing and | positivity. | positivity | exercise, group |
| reframing negative thoughts and | 2. Daily gratitude habits (3 Good | checklist, | brainstorm, gratitude |
| fostering optimistic thinking | Things Journal). | gratitude | journaling, resilience |
| habits | 3. Practice of resilience (self- | journal | sharing, mood |
| | awareness, social support, | worksheets. | tracking tools. |
| | meaning, optimism). | | |
| | 4. Activities to build resilience | | |
| | (Small Wins Journal, Self-Talk | | |
| | Assessment, Brief Resilience | | |
| | Scale). | | |
| | 5. Role-playing to reframe | | |
| | negative thoughts (e.g., handling | | |
| | family complaints). | | |
| | 6. Progressive muscle relaxation | | |
| | (5-10 min) paired with gratitude | | |
| | journaling. | | |
| Session 4: Tea | mwork and Well-being in Paedia | tric Oncology N | Nursing |
| Objective | Content (Topics) | Materials/Aids | Teaching strategy |
| Objective Recognize individual roles in | ` | Materials/Aids<br>Teamwork | Teaching strategy Thought Reframing |
| Ü | ` | | |
| Recognize individual roles in | 1. The Strength of Teamwork | Teamwork | Thought Reframing |
| Recognize individual roles in patient outcomes, build team | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect</li> </ol> | Teamwork reflection | Thought Reframing Exercise, Group |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect</li> </ol> | Teamwork<br>reflection<br>sheets, trust- | Thought Reframing Exercise, Group Brainstorm, Gratitude |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect</li> </ol> | Teamwork<br>reflection<br>sheets, trust-<br>building | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress | The Strength of Teamwork Building Trust and Respect within Teams: | Teamwork reflection sheets, trust- building activity | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing Teams</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict resolution | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving exercise, team |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing Teams</li> <li>Setting Boundaries to Protect</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict resolution | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving exercise, team reflection activity, |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress reduction. | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing Teams</li> <li>Setting Boundaries to Protect</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict resolution | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving exercise, team reflection activity, |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress reduction. | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing Teams</li> <li>Setting Boundaries to Protect Personal Time</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict resolution | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving exercise, team reflection activity, |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress reduction. | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing Teams</li> <li>Setting Boundaries to Protect Personal Time</li> <li>Developing a Personal Follow-up Plan</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict resolution | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving exercise, team reflection activity, |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress reduction. | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing Teams</li> <li>Setting Boundaries to Protect Personal Time</li> <li>Developing a Personal Follow-up Plan</li> <li>Effective Communication</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict resolution | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving exercise, team reflection activity, |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress reduction. | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing Teams</li> <li>Setting Boundaries to Protect Personal Time</li> <li>Developing a Personal Follow-up Plan</li> <li>Effective Communication Skills: Connecting with Empathy:</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict resolution | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving exercise, team reflection activity, |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress reduction. | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing Teams</li> <li>Setting Boundaries to Protect Personal Time</li> <li>Developing a Personal Follow-up Plan</li> <li>Effective Communication Skills: Connecting with Empathy: <ul> <li>Active listening and empathy.</li> </ul> </li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict resolution | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving exercise, team reflection activity, |
| Recognize individual roles in patient outcomes, build team unity through trust and respect, and advocate for systemic stress reduction. | <ol> <li>The Strength of Teamwork</li> <li>Building Trust and Respect within Teams:</li> <li>Problem Solving in Nursing Teams</li> <li>Setting Boundaries to Protect Personal Time</li> <li>Developing a Personal Follow-up Plan</li> <li>Effective Communication Skills: Connecting with Empathy:</li> </ol> | Teamwork reflection sheets, trust- building activity instructions, conflict resolution | Thought Reframing Exercise, Group Brainstorm, Gratitude Journaling, Resilience Sharing, Mood Tracking Tools. Problem-solving exercise, team reflection activity, |

### Session1: Self-Care for Nurses: Managing Occupational Stress and Preventing Burnout

### 1 Introduction (10 minutes)

This teaching guide provides detailed instructions for facilitating Session 1 of the Nurses' Stress Self-Care Educational Program, designed for paediatric oncology nurses in selected Jordanian hospitals. The session introduces the study, its purpose, risks, benefits, and activities, emphasizing a culturally relevant initiative for professional and personal growth. The programme aims to assist nurses in managing burnout and occupational stress, with a structure spanning three days over two weeks, including two two-hour sessions and a one-hour follow-up session. A one-month booster session and a peer support WhatsApp group will sustain engagement.

- 1. Study Overview (5 minutes): Introduce the study, explaining its purpose to improve nurses' self-care management of burnout and occupational stress. Highlight that it is part of a doctoral degree requirement, with no known risks based on prior studies. Emphasize voluntary participation, confidentiality (using three-digit codes, e.g., I-A-1 for intervention group, hospital A, participant 1), and no penalties for non-participation. Mention certificates of participation upon completion.
- **2.** Consent and Questionnaires (3 minutes): Guide participants to sign the Informed Consent Form. Explain the questionnaires, ensuring clarity on each item, and address any questions. Outline the data collection process (pre-workshop, post-workshop, and one-month follow-up) to ensure accuracy.
- **3. Programme Structure** (**2 minutes**): Describe the workshop structure: three days over two weeks, with two two-hour sessions and a one-hour follow-up session arranged with the nursing manager. Introduce the one-month booster session and WhatsApp group for peer support.

### **2** Workshop Objectives (10 minutes)

### 2.1 Overview

This segment outlines the objectives of the workshop, focusing on equipping nurses with practical skills to differentiate stress from burnout, identify workplace stressors, develop self-care strategies, create a burnout prevention plan, and advocate for systemic changes in Jordanian hospitals.

### 2.2 Facilitation Steps

- 1. Interactive Lecture (5 minutes): Present the objectives using a flip chart:
  - Differentiate between healthy stress and burnout.
  - Identify sources of stress in the nursing work environment.
  - Learn practical skills for psychological self-care and daily stress management.
  - Develop a personal and realistic burnout prevention plan.
  - Advocate for systemic changes to reduce workplace stress in Jordanian hospitals.
- **2. Group Discussion (5 minutes)**: Facilitate a brief discussion asking participants to share one personal goal for the workshop related to stress management. Record key points on the flip chart to build engagement.

### **3** Key Definitions of Occupational Stress and Burnout (15 minutes)

### 3.1 Overview

This segment defines occupational stress and burnout, highlighting common sources and symptoms relevant to paediatric oncology nurses, supported by WHO and Maslach's frameworks.

- 1. **Definitions and Sources (7 minutes)**: Use an interactive lecture to define occupational stress (WHO, 2021: a psychological and physiological response when job demands exceed capacity) and burnout (Maslach & Leiter, 2016: chronic stress with emotional exhaustion, depersonalization, and reduced personal accomplishment). List common sources on a flip chart: limited resources, high workload, job insecurity, conflicts, violence, staff shortages, difficult relationships, verbal/physical abuse, equipment shortages, night shifts, and lack of support.
- **2. Symptoms Table (5 minutes)**: Display Table 1 (Occupational Stress Common Symptoms) using a handout or flip chart:
- **3. Reflection (3 minutes)**: Ask participants to identify one symptom they've experienced and write it on their reflection worksheets, discussing its impact briefly in pairs.

**Table (1): Occupational stress common symptoms** 

| Physical signs | Mental signs |
|---|---|
| Fast heartbeat | Difficulty concentrating |
| <ul> <li>Breathing Difficulties</li> </ul> | <ul> <li>Obsessing on the situation</li> </ul> |
| Headache | <ul> <li>Revenge thoughts</li> </ul> |
| <ul> <li>Stomach discomfort</li> </ul> | <ul> <li>Negative thinking</li> </ul> |
| <ul> <li>Sweating</li> </ul> | |
| <ul> <li>Feeling hot in the face or neck</li> </ul> | |
| Trembling | |
| Emotional signs | Behavioural signs |
| Emotional signs Sadness | Behavioural signs Clenched fists |
| | Ö |
| • Sadness | Clenched fists |
| <ul><li>Sadness</li><li>Irritability</li></ul> | <ul><li>Clenched fists</li><li>Pounding of fist on any surface</li></ul> |
| <ul><li>Sadness</li><li>Irritability</li><li>Guilt</li></ul> | <ul> <li>Clenched fists</li> <li>Pounding of fist on any surface</li> <li>Pacing</li> </ul> |
| <ul> <li>Sadness</li> <li>Irritability</li> <li>Guilt</li> <li>Resentment</li> </ul> | <ul> <li>Clenched fists</li> <li>Pounding of fist on any surface</li> <li>Pacing</li> <li>Raising one's voice</li> </ul> |

### **4** Effects of Stress on the Body and Mind (15 minutes)

### 4.1 Overview

This segment explores the short-term and long-term effects of stress on nurses physical and mental health, emphasizing the progression from early symptoms to chronic conditions if stressors persist.

- **1. Lecture on Stress Effects (7 minutes)**: Explain short-term stress (immediate physical responses) versus long-term stress (chronic health issues). Present Table 2 (Occupational Stress Related Problems) on a flip chart or handout:
- **2. Group Activity (5 minutes)**: Facilitate a group brainstorm on one short-term and one long-term effect they have noticed in their work environment. Write responses on the flip chart.
- **3. Reflection (3 minutes)**: Ask participants to write one stress effect they have experienced and a potential coping strategy on their reflection worksheets.

**Table (2): Occupational stress related problems** 

| | Early Physical Symptoms | Early Mental signs |
|-------|------------------------------|--------------------------------------|
| | Headaches | > Anxiety |
| _ | Digestive issues | Irritability or mood swings |
| Term | Eating disturbances | Low morale |
| | Sleep disturbances | Depression |
| ort | Fatigue | Alcohol & drug use |
| Short | Muscle aches & pains | Feeling powerless |
| | Frequent minor illnesses | Isolation from co- workers. |
| | Chronic Physical Conditions* | Psychological & Behavioral Problems* |
| | High Blood Pressure | Serious depression |
| _ | Heart disease | Suicidal behavior |
| erm | Stroke | Domestic violence |
| Te | Spastic colon | Alcohol abuse |
| gu | Immune system dysfunction | Substance abuse |
| Long | Diabetes | Burnout. |
| | Asthma | |
| | Musculoskeletal disorders. | |

<sup>\*</sup> If exposure to stressors continues for a longer period of time, chronic health problems can develop

### 5 The Importance of Self Stress Management Programme (10 minutes)

### 5.1 Overview

This segment emphasizes the benefits of effective stress management for nurses health, job satisfaction, and patient care quality, introducing problem-focused and emotion-focused coping strategies.

- **1. Interactive Lecture (5 minutes)**: Discuss how stress management improves nurse health, care quality, and institutional outcomes. Introduce coping strategies (Figure 1):
  - **Problem-focused coping**: Aims to change/remove stress causes (e.g., seeking solutions, setting boundaries, planning).
  - Emotion-focused coping: Manages uncomfortable feelings (e.g., talking and rest)
- **2. Paired Discussion (3 minutes)**: Pair participants to share one example of a coping strategy they have used (problem- or emotion-focused). Distribute communication skill checklists to guide interactions.
- **3. Reflection (2 minutes)**: Ask participants to write one coping strategy they will try this week on their reflection worksheets.



Figure (1): Coping Strategies Types

### **6** Notes for Facilitators

- Create a safe, non-judgmental environment to encourage open sharing, critical for effective discussions.
- Monitor time closely to cover all segments within the 1-hour session.
- Use examples relevant to paediatric oncology nursing (e.g., high workload, emotional patient interactions) to make activities relatable.
- Ensure all participants have access to reflection worksheets and communication skill checklists.
- Adapt discussions to group dynamics, offering alternative scenarios if needed.

### Session 2: Nurture Interpersonal Connections – Building Your Support Network

### 1 Detailed Content and Facilitation

### 1.1 Stress Management Techniques (20 minutes)

### 1.1.1 Overview

This segment introduces evidence-based tools to manage stress, including deep breathing, progressive muscle relaxation, time management, and grounding techniques, which reduce physiological and psychological stress in healthcare professionals.

### 1.1.2 Facilitation Steps

**1. Introduction (3 minutes)**: Explain the importance of stress management for nurses, noting its impact on reducing cortisol levels and improving well-being. Use the flip chart to write key terms: "Deep Breathing," "Progressive Muscle Relaxation," "Time Management," and "Grounding Techniques."

### 2. Deep Breathing Exercise (5 minutes):

- Guide participants through a 4-7-8 breathing exercise: Inhale for 4 seconds, hold for 7 seconds, exhale for 8 seconds, as supported by research on diaphragmatic breathing for stress reduction.
- Demonstrate first, then lead the group through 3 rounds.
- Encourage participants to note how they feel in their reflection worksheets.

### 3. Progressive Muscle Relaxation (5 minutes):

- Instruct participants to tense and relax muscle groups (e.g., hands, shoulders, legs) for 5 seconds each, following established protocols.
- Lead a 5-minute session, focusing on major muscle groups.
- Ask participants to record observations in their reflection worksheets.

### 4. Time Management Skills (4 minutes):

- Discuss prioritization and delegation using the Eisenhower Matrix, a proven time management tool.
- Encourage paired discussion: Share one-time management challenge and a potential solution.

### 5. Grounding Techniques (3 minutes):

- Introduce the 5-4-3-2-1 technique: Identify 5 things you see, 4 you can touch, 3 you hear, 2 you smell, 1 you taste, effective for anxiety reduction.
- Lead a brief practice and discuss its application during stressful shifts.

### 1.2 Resilience Training (20 minutes)

### 1.2.1 Overview

This segment focuses on building long-term resilience through optimism, problem-solving, support networks, and finding meaning and purpose, which are critical for mitigating burnout in nurses.

### 1.2.2 Facilitation Steps

### 1. Developing an Optimistic Outlook (5 minutes):

- Use an interactive lecture to discuss optimism as a resilience factor, which can reduce burnout symptoms.
- Example: Share a short story of a nurse who reframed a challenging shift positively.
- Ask participants to write one optimistic thought about their work on their reflection worksheets.

### 2. Problem-Solving Skills (5 minutes):

- Introduce a simple problem-solving framework (e.g., Identify, Analyse, Plan, Act), supported by research on structured problem-solving in clinical settings.
- Use a flip chart to outline a nursing scenario (e.g., managing a heavy patient load).
- Facilitate a group discussion to brainstorm solutions.

### 3. Building a Support Network (5 minutes):

- Discuss the value of peer support in nursing, which significantly reduces stress and enhances coping.
- Pair participants for a 2-minute listening exercise: One shares a workplace challenge, the other listens actively without interrupting.
- Distribute communication skill checklists to guide future interactions.

### 4. Finding Meaning and Purpose (5 minutes):

- Discuss the spiritual rewards of nursing, such as impacting lives, which enhances resilience and job satisfaction.
- Introduce "purpose mapping." Participants write one daily task and connect it to a core value (e.g., compassion, service) on their reflection worksheets.
- Encourage sharing in small groups to reinforce purpose-driven work.

### **1.3** Self-Compassion Practices (10 minutes)

### 1.3.1 Overview

This segment teaches participants to practice self-compassion, which reduces burnout by fostering kindness toward oneself and recognizing shared human experiences.

### 1.3.2 Facilitation Steps

**1. Introduction (2 minutes)**: Explain self-compassion using the three elements: self-kindness, common humanity, and mindfulness, as outlined by Neff.

### 2. Empathy Role-Play (6 minutes):

- Have participants role-play a scenario where one nurse feels overwhelmed and the other offers self-compassionate responses (e.g., "It's okay to feel this way, you're not alone").
- Use the communication skill checklist to guide responses.
- **3. Reflection (3 minutes)**: Ask participants to write a self-compassionate message to themselves on their reflection worksheets, addressing a recent challenge.

### 1.4 Cognitive Restructuring (10 minutes)

### 1.4.1 Overview

This segment introduces Cognitive Behavioural Therapy (CBT)-based techniques to identify and challenge negative thought patterns, replacing them with positive ones to manage stress effectively.

### 1.4.2 Facilitation Steps

1. Introduction (3 minutes): Explain cognitive restructuring using a flip chart to illustrate the process: Identify negative thought → Challenge it → Replace with a positive thought, as described in CBT literature.

### 2. Group Activity (5 minutes):

- Provide a common negative thought (e.g., "I'm not good enough for this job").
- Facilitate a group brainstorm to challenge and reframe it (e.g., "I'm learning and improving every day").
- Write responses on the flip chart.
- **3. Reflection (2 minutes)**: Ask participants to identify one negative thought from their workweek and write a reframed version on their reflection worksheets.

### **2** Wrap-Up and Mentorship Planning (10 minutes)

**1. Group Discussion (5 minutes)**: Facilitate a discussion on key takeaways from the session. Ask: "What's one technique you'll try this week?"

### 2. Mentorship Planning (5 minutes):

- Encourage participants to form mentorship pairs for ongoing support, as peer support enhances resilience and reduces burnout.
- Distribute reflection worksheets with a section for planning weekly check-ins with a mentor or peer.
- Emphasize using communication skills (from the checklist) in mentorship.

### **3** Notes for Facilitators

- Create a safe, non-judgmental environment to encourage open sharing, which is critical for effective group discussions.
- Monitor time closely to cover all segments within the 1-hour session.
- Be prepared to offer examples relevant to nursing (e.g., patient care challenges) to make activities relatable.
- Ensure all participants have access to reflection worksheets and communication skill checklists.
- Adapt role-plays to the group's dynamics, offering alternative scenarios if needed.

### **Session 3: Reframing Stressful Thoughts with Positive Thinking**

### 1 Develop an Attitude of Positivity Cultivating Hope and Resilience (20 minutes)

### 1.1 Overview

This segment introduces positive thinking as a tool to enhance resilience and problem-solving under stress, particularly for paediatric oncology nurses in Jordanian hospitals. It focuses on identifying and counteracting negative thinking patterns (catastrophizing, overgeneralizing, personalizing, filtering) and implementing six steps to foster positive self-talk, which can improve energy, control, and purposeful action.

- 1. Interactive Lecture (5 minutes): Explain how positive thinking helps nurses feel better, stay resilient, and solve problems effectively. Define negative thinking patterns (catastrophizing, overgeneralizing, personalizing, filtering) using a flip chart. Highlight the importance of positive self-talk for managing stress and enhancing growth.
- **2. Eliminate Internal Negative Chatter (3 minutes)**: Discuss the need for awareness of negative thoughts. Lead a brief exercise where participants identify one negative thought they have had recently (e.g., I can't handle this shift). Ask them to write it on their reflection worksheets and note its impact on their mood.
- **3. Positive Affirmations (3 minutes)**: Introduce affirmations as short, believable statements repeated daily to rewire thinking. Provide examples (e.g., I am capable of managing challenges). Guide participants to write one affirmation on their reflection worksheets and practice saying it aloud.
- **4. Positive Scripts (4 minutes)**: Present positive mental scripts (e.g., Calm down first, and think this through, I am capable of managing this situation). Display the list on a flip chart. Facilitate a paired discussion where participants share one script they could use during a stressful shift.
- **5. Replace Negative Influences with Positive Ones (3 minutes)**: Discuss identifying external negative influences (e.g., unsupportive colleagues). Encourage participants to brainstorm one positive influence (e.g., a supportive mentor) and write it on their reflection worksheets.
- **6.** Confront Fears and Focus on Enjoyable Moments (2 minutes): Explain how confronting fears and focusing on positive moments builds resilience. Lead a brief group discussion on one enjoyable moment from their workweek to shift focus to positivity.

### 2 Daily Gratitude Habit (3 Good Things Journal) (10 minutes)

### 2.1 Overview

This segment teaches the practice of gratitude to shift focus from deficits to positive aspects of life, reducing stress and enhancing well-being among nurses. Writing three things they are thankful for daily fosters positive emotions.

### 2.2 Facilitation Steps

- **1. Introduction (3 minutes)**: Explain the benefits of gratitude for mental health and stress reduction, supported by research. Use a flip chart to write 3 Good Things Journal and describe the practice of noting three daily things to be thankful for.
- **2. Group Activity (4 minutes)**: Guide participants to write three things they are grateful for from the past week on their reflection worksheets (e.g., a kind patient interaction, a supportive colleague). Facilitate a brief sharing in small groups to reinforce positivity.
- **3. Reflection (3 minutes)**: Ask participants to commit to practicing the 3 Good Things Journal daily for a week and write a plan for integrating it into their routine on their reflection worksheets.

### **3** Practice of Resilience (15 minutes)

### 3.1 Overview

This segment focuses on building resilience among paediatric oncology nurses through self-awareness, social support, meaning and purpose, and realistic optimism, which enhance job satisfaction and patient outcomes.

### 3.2 Facilitation Steps

**1. Lecture on Resilience Components (5 minutes)**: Present Table 5 (Core Components of Resilience) on a flip chart or handout:

**Table (5): Core Components of Resilience** 

| <b>Resilience Components</b> | Descriptions |
|---|---|
| 1. Self-awareness | Know how you react to stress |
| | <b>Example:</b> Notice when you're emotionally triggered and why |
| 2. Social support | Trusted relationships reduce pressure |
| | <b>Example:</b> Regular debriefing with a fellow nurse |
| 3. Meaning and purpose | Connect daily tasks to personal values |
| | <b>Example:</b> "I'm doing this because I believe every child |
| | deserves dignity" |
| 4. Realistic optimism | Focus on what you can control |
| | <b>Example:</b> "I can't fix staffing, but I can ask for help" |

- **2. Group Discussion (5 minutes)**: Facilitate a discussion on one resilience component participants find most relevant. Ask them to share an example from their work (e.g., a moment of self-awareness or seeking support).
- **3. Reflection (5 minutes)**: Ask participants to select one component and write a plan to strengthen it (e.g., scheduling a debrief with a colleague) on their reflection worksheets.

### 4 Activities to Build Resilience (15 minutes)

### 4.1 Overview

This segment provides practical activities to reinforce resilience through journaling, self-talk assessment, a resilience scale, and role-playing, tailored to the challenges faced by paediatric oncology nurses.

### **4.2** Facilitation Steps

- **1. Small Wins Journal (3 minutes)**: Introduce the Small Wins Journal, where participants write three things they did well each week. Guide them to start with one example on their reflection worksheets to build self-efficacy.
- **2. Self-Talk Assessment (4 minutes)**: Distribute a handout with the Self-Talk Assessment checklist:
  - I notice that I criticize myself a lot.
  - I say to myself phrases like I can't or I always fail.
  - I try to change these phrases to more encouraging ones.
  - I use positive phrases when I face a difficult situation.
  - I talk to myself like I would talk to a friend going through a difficult situation.

Ask participants to check applicable statements and discuss one in pairs.

- **3. Brief Resilience Scale (BRS) (3 minutes)**: Explain the 6-item BRS as a tool to assess resilience. Guide participants to complete it on their reflection worksheets and reflect on one area for growth, not as a label.
- **4. Role-Playing (5 minutes)**: Facilitate a role-play scenario (e.g., handling family complaints in a Jordanian hospital). One nurse expresses a negative thought, and the other reframes it positively. Follow with a brief point-based quiz to reinforce learning, using the communication skill checklist.

### **5** Notes for Facilitators

- Create a safe, non-judgmental environment to encourage open sharing, critical for effective discussions.
- Monitor time closely to cover all segments within the 1-hour session.
- Use examples relevant to paediatric oncology nursing (e.g., emotional patient interactions, family complaints) to make activities relatable.
- Ensure all participants have access to reflection worksheets and communication skill checklists.
- Adapt role-plays to group dynamics, offering alternative scenarios if needed.

### Session 4: Teamwork and Well-being in Paediatric Oncology Nursing

### 1 The Strength of Teamwork (10 minutes)

### 1.1 Overview

This segment highlights the importance of effective teamwork in paediatric oncology nursing for delivering high-quality care and reducing occupational stress and burnout. It emphasizes the multidisciplinary nature of teams and the critical role of each nurses skills, knowledge, and compassion in improving patient outcomes and fostering team resilience.

### 1.2 Facilitation Steps

- **1. Interactive Lecture (5 minutes)**: Explain the role of multidisciplinary teams (oncologists, nurses, sociologists, dietitians) in paediatric oncology, focusing on shared goals, face-to-face interactions, and improved patient welfare. Use a flip chart to list key points: shared identity, nurse contributions, and impact on stress reduction.
- **2. Group Discussion (3 minutes)**: Facilitate a discussion asking participants to share one example of how their contribution (e.g., compassion, attention to detail) impacted a patient or family. Record key points on the flip chart to reinforce pride and responsibility.
- **3. Reflection (2 minutes)**: Ask participants to write one strength they bring to their team on their reflection worksheets, emphasizing its role in patient care and team resilience.

### **2** Building Trust and Respect within Teams (15 minutes)

### 2.1 Overview

This segment focuses on fostering a supportive environment through respect and conflict resolution, critical for teamwork in high-pressure paediatric oncology units. It introduces techniques like active listening, open communication, mutual respect, reliability, and empathy to enhance team cohesion.

- 1. Lecture on Trust and Respect (5 minutes): Present the importance of respect and conflict resolution in teams. Use a flip chart to list techniques: active listening, open communication, mutual respect, reliability, and empathy. Explain their role in reducing stress and improving care quality.
- **2. Paired Activity (5 minutes)**: Pair participants for a 2-minute active listening exercise: one shares a workplace challenge, the other practices active listening (nodding, eye contact, no interrupting). Distribute communication skill checklists to guide interactions.
- **3. Group Discussion (5 minutes)**: Facilitate a discussion on one technique (e.g., empathy) participants find valuable. Ask them to share an example of applying it in their team. Write responses on the flip chart.

### **3** Problem Solving in Nursing Teams (15 minutes)

### 3.1 Overview

This segment introduces team-based problem-solving as a core skill in nursing, using a structured six-step process to address barriers (e.g., delayed medication delivery) while fostering trust and safe care.

### 3.2 Facilitation Steps

**1. Lecture on Problem-Solving Steps (5 minutes)**: Present Table 6 (Problem Solving Steps) on a flip chart or handout:

**Table (6): Problem Solving Steps** 

| Step | Actions |
|---|---|
| 1. Identify the Problem | Describe it clearly, involve others: |
| | Ask: What exactly is wrong? |
| | • Is it a one-time issue or does it happen often? |
| | Involve others to describe the problem clearly |
| | Tip: Don't rush. A wrong diagnosis of the problem wastes time |
| 2. Understand the Problem | Gather facts, see full impact: |
| | Collect facts, not opinions |
| | Observe how the issue affects workflow or patient care |
| | <ul> <li>Include all voices: nurses, physicians, support staff</li> </ul> |
| | Goal: See the full picture before jumping to solutions |
| 3. Suggest Solutions | Brainstorm as a team: |
| | Avoid judging ideas too early |
| | Encourage everyone to speak |
| | Good example: Create a new handover checklist if critical information |
| | is missed |
| 4. Decide on a Solution | Choose what works, consider risks: |
| | Evaluate the options |
| | Which is doable with your resources? |
| | What will cause the least disruption? |
| | • Important: Always consider "What happens if we do nothing?" |
| 5. Act | Assign tasks, stay flexible |
| | Assign clear roles |
| | Communicate the plan |
| | Document what you're doing The Grand Hard State of the Control of the Contr |
| | Tip: Stay flexible. Be ready to adjust if new problems appear |
| 6. Follow Up | Evaluate, adjust, and share learning |
| | • Did the solution work? |
| | Get feedback from team members and patients To all the the relationships and patients. |
| | Track whether the issue repeats |
| | Share results so everyone learns |

- **2. Group Activity** (**7 minutes**): Present a scenario (e.g., delayed chemotherapy medication). Facilitate a group brainstorm to apply the six steps, writing solutions on the flip chart. Emphasize including all voices and avoiding blame.
- **3. Reflection (3 minutes)**: Ask participants to write one problem-solving step they will apply in their next team challenge on their reflection worksheets.

### **4** Setting Boundaries to Protect Personal Time (10 minutes)

### 4.1 Overview

This segment teaches strategies to set boundaries in the demanding paediatric oncology field to prevent burnout and preserve personal well-being, tailored to Jordanian nurses work environment.

### 4.2 Facilitation Steps

- **1. Introduction (3 minutes)**: Explain the importance of boundaries to protect personal time. Use a flip chart to list strategies: know your limits, prioritize needs, communicate assertively, practice saying no, establish no work zones, seek support.
- **2. Paired Discussion** (**4 minutes**): Pair participants to share one boundary-setting challenge (e.g., work calls on days off) and a potential strategy. Use communication skill checklists to guide assertive communication.
- **3. Reflection (3 minutes)**: Ask participants to write one boundary they will set this week (e.g., no work emails after 7 PM) on their reflection worksheets.

### 5 Developing a Personal Follow-up Plan (10 minutes)

### 5.1 Overview

This segment guides nurses in creating a personal follow-up plan to sustain stress management and resilience, using self-assessment, skill practice, peer check-ins, progress logging, and re-evaluation.

### **5.2** Facilitation Steps

**1. Lecture on Follow-up Plan (4 minutes)**: Present the follow-up plan components using a flip chart: weekly self-assessment, skill practice, peer check-ins, logging progress, two-month re-evaluation. Display the Sample Follow-up Plan Template:

### **Sample Follow-up Plan Template**

| How to Track Progress | Time | Description | Activity |
|---|---|---|---|
| Use a digital or paper log | Friday | Rate stress and resilience levels | Weekly Check – in |
| Mark on a calendar | Morning | 5 Minute daily exercise | Deep Breathing |
| Short bullet notes after talk | Thursday | 10 Minutes weekly conversation | Partner Reflection |
| Compare with initial scores | After 8 weeks | Fill burnout / resilience scale | 2 Month Evaluation |

- **2. Group Activity (4 minutes)**: Guide participants to draft one part of their follow-up plan (e.g., choosing a weekly skill like positive affirmations) on their reflection worksheets. Facilitate brief sharing in small groups.
- **3. Reflection (2 minutes)**: Ask participants to commit to one follow-up action (e.g., weekly stress rating) and write it on their reflection worksheets.

### **6** Effective Communication Skills: Connecting with Empathy (10 minutes)

### 6.1 Overview

This segment emphasizes empathy and active listening to prevent burnout and enhance team cohesion in paediatric oncology nursing, aligning with Jordanian cultural values of strong interpersonal relationships.

### **6.2** Facilitation Steps

- **1. Lecture on Communication Skills (3 minutes)**: Explain how empathy and active listening reduce stress and build trust. List skills on a flip chart: active listening, empathy, nonverbal cues, clarity, and feedback. Note the cultural relevance in Jordanian settings [2].
- **2. Video and Discussion (5 minutes)**: Show a 2-minute video on assertiveness in nursing (https://www.youtube.com/watch?v=hEKrJj\_0DU4). Facilitate a brief discussion on how empathy applies to patient and team interactions. Use communication skill checklists to guide responses.
- **3. Reflection (2 minutes)**: Ask participants to write one communication skill they will practice (e.g., summarizing a colleagues concern) on their reflection worksheets.

### 7 Active Listening and Empathy (10 minutes)

### 7.1 Overview

This segment explores active listening and empathetic listening as tools to enhance communication, using dimensions of listening and Coveys empathetic listening tasks to foster under- standing in high-stress settings.

### 7.2 Facilitation Steps

**1. Lecture on Listening Dimensions (4 minutes)**: Present Table 7 (Active Listening Dimension) on a flip chart or handout:

**Table 7: Active Listening Dimension** 

| Dimension | Description |
|---|---|
| The occasion for the message | What is the reason why the person is communicating with me now? |
| The length of the message | What can the length of the message tell me about its importance? |
| The words chosen | Is the message being made formally? Is it with aloofness or slang? |
| The volume and pace | What clues do the loudness and speed give me? |
| The Pauses and Hesitations | How do these enhance or detract from the message? |
| Non-verbal clues | What does eye contact, posture, or facial expressions tell me about the message? |

Explain Coveys five empathetic listening tasks: repeat verbatim, rephrase content, reflect feelings, combine content and feelings, discern when empathy is not needed.

- **2. Paired Role-Play (4 minutes)**: Pair participants to practice empathetic listening: one shares a patient interaction challenge, the other applies one listening task (e.g., reflecting feelings). Use communication skill checklists
  - **8** The Power of Non-Verbal Communication (5 minutes)

### 8.1 Overview

This segment highlights the impact of non-verbal communication (body language, gestures) on effective interactions, noting its significant role in conveying emotions in nursing.

- (a) Introduction (3 minutes): Explain non-verbal communications role (93
- (b) **Group Activity (2 minutes)**: Facilitate a quick exercise where participants practice positive body language (e.g., open posture, eye contact) in pairs, noting its effect on communication.

### 9 Strategic Questioning as a Tool in Active Listening (5 minutes)

### 9.1 Overview

This segment teaches active questioning techniques (open-ended, clarifying, closed, reflective) to enhance communication and understanding in nursing interactions.

- (a) **Lecture on Questioning Types (3 minutes)**: Present Table 8 (Active Questioning) on a flip chart or handout:
- (b) **Reflection (2 minutes)**: Ask participants to write one questioning type they will use in their next patient or colleague interaction on their reflection worksheets

**Table (8): Active Questioning** 

| Question type | Description |
|---|---|
| Open ended Questions | Open questions stimulate thinking and discussion or responses including |
| | opinions or feelings. They pass control of the conversation to the respondent. |
| | Leading words in open questions include: Why, what, or how, as in the |
| | following examples: |
| | Could you tell me more shout the pain you've been experiencine? |
| | Could you tell me more about the pain you've been experiencing? How have you been feeling since your last medication change? |
| | How did that make you feel? |
| <b>Clarifying Questions</b> | A clarifying question helps to remove ambiguity, elicits additional detail, and guides the answer to a question. When you ask a clarifying question, you ask |
| | for expansion or detail, while withholding your judgment and own opinions. When asking for clarification, you will have to listen carefully to what the other |
| | person says. Frame your question as someone trying to understand in more detail. Often asking for a specific example is useful. This also helps the speaker evaluate his or her own opinions and perspective. Below are some examples: |
| | Example (1): Can you explain more about that moment? |
| | Example (2): Patient says: "I've just been feeling really off lately." Nurse asks: "Could you tell me more about what you mean by 'off'? For example, have you noticed any changes in your energy levels, appetite, or sleep?" |
| | Example (3): Patient says: "This medication isn't working." |
| | <b>Nurse asks:</b> "Can you describe what you've noticed that makes you say it isn't working? Are your symptoms staying the same, getting worse, or are you experiencing new side effects?" |
| <b>Closed Questions</b> | Closed questions usually require a one-word answer, and effectively shut off |
| | discussion. Closed questions provide facts, allow the questioner to maintain |
| | control of the conversation, and are easy to answer. Typical leading words are: |
| | Is, can, how many, or does. While closed questions are not the optimum choice for active listening, at times they may be necessary to elicit facts. Below are several examples of closed questions: |
| | Are you experiencing any pain right now? |
| | Have you taken your medication this morning? |
| Reflective | You seem worried—did I understand right? |
| i | |

### **10** Notes for Facilitators

- Create a safe, non-judgmental environment to encourage open sharing, critical for effective discussions.
- Monitor time closely to cover all segments within the 1-hour session.
- Use examples relevant to paediatric oncology nursing (e.g., patient family interactions, medication delays) to make activities relatable.
- Ensure all participants have access to reflection worksheets and communication skill checklists.
- Adapt role-plays and discussions to group dynamics, offering alternative scenarios if needed.

**Conclusion: Sustaining Your Compassion Journey** 

Dear Paediatric Oncology Nurse,

This manual has provided a framework to recognise and control burnout through focusing on

finding meaning, nurturing your inner resources, building strong connections, cultivating

positivity, and prioritising your overall well-being. Remember that burnout prevention and

self-care are ongoing processes, not destinations.

We encourage you to revisit these concepts and practices regularly. Integrate the strategies that

resonate most with you into your daily life, both personally and professionally. When you need

support, seek it out, and remember the profound impact on the lives of your patients and their

families.

Your work is invaluable and there are instances of good. By prioritising your own care, you

protect not only yourself but also enhance your ability to provide good and sustainable care for

the children who need you the most. You can find constant strength, purpose, and joy in your

extraordinary vocation.

Thank you for your unwavering dedication, your compassionate hearts, and your tireless efforts

in the field of paediatric oncology nursing. Your work makes a world of difference.

24

### **References and reading Materials**

Ano, G. G., & Vasconcelles, E. B. (2005). Religious coping and psychological adjustment to stress: A meta-analysis. *Journal of Clinical Psychology*, 61(4), 461–480. https://doi.org/10.1002/jclp.20049

Folkman, S., & Moskowitz, J. T. (2004). Coping: Pitfalls and promise. *Annual Review of Psychology*, 55, 745–774. https://doi.org/10.1146/annurev.psych.55.090902.141456

Maslach, C., & Leiter, M. P. (2016). Understanding the burnout experience: Recent research and its implications for psychiatry. *World Psychiatry*, *15*(2), 103–111. <a href="https://doi.org/10.1002/wps.20311">https://doi.org/10.1002/wps.20311</a>

Mealer, M., Jones, J., & Moss, M. (2012). A qualitative study of resilience and posttraumatic stress disorder in United States ICU nurses. *Intensive Care Medicine*, *38*(9), 1445–1451. https://doi.org/10.1007/s00134-012-2600-6

Neff, K. D. (2003). Self-compassion: An alternative conceptualization of a healthy attitude toward oneself. *Self and Identity*, 2(2), 85–101. <a href="https://doi.org/10.1080/15298860309032">https://doi.org/10.1080/15298860309032</a>

Nopa, I., Kurniawidjaja, L. M., Erwandi, D. J. C. S. P. J. o. P. H., & Health, C. (2023). Religious Coping Strategies For Nurses' Work Related Stress: A Scoping Review. 5(2), 435-450. https://doi.org/10.30829/contagion.v5i2.15197

O'Daniel, M., & Rosenstein, A. H. (2008). Professional communication and team collaboration. In R. G. Hughes (Ed.), *Patient safety and quality: An evidence-based handbook for nurses* (pp. 2–271–2–284). Agency for Healthcare Research and Quality. <a href="https://www.ncbi.nlm.nih.gov/books/NBK2637/">https://www.ncbi.nlm.nih.gov/books/NBK2637/</a>

Park, C. L. (2010). Making sense of the meaning literature: An integrative review of meaning making and its effects on adjustment to stressful life events. *Psychological Bulletin*, *136*(2), 257–301. <a href="https://doi.org/10.1037/a0018301">https://doi.org/10.1037/a0018301</a>

Parks, L. (2021). *Unifying Vision: Strategies that Influence Nurse Self-Care Practices in Intensive Care Unit Nurses*. https://digitalcommons.jsu.edu/etds\_nursing/44/

Pargament, K. I. (1997). The psychology of religion and coping: Theory, research, practice. Guilford Press.

Salas, E., Sims, D. E., & Burke, C. S. (2005). Is there a "Big Five" in teamwork? *Small Group Research*, *36*(5), 555–599. <a href="https://doi.org/10.1177/1046496405277134">https://doi.org/10.1177/1046496405277134</a>

- Shanafelt, T. D., & Noseworthy, J. H. (2017). Executive leadership and physician well-being: Nine organizational strategies to promote engagement and reduce burnout. *Mayo Clinic Proceedings*, 92(1), 129–146. https://doi.org/10.1016/j.mayocp.2016.10.004
- Smith, B. W., Dalen, J., Wiggins, K., Tooley, E., Christopher, P., & Bernard, J. (2008). The brief resilience scale: Assessing the ability to bounce back. *International Journal of Behavioral Medicine*, 15(3), 194–200. https://doi.org/10.1080/10705500802222972
- Tugade, M. M., & Fredrickson, B. L. (2004). Resilient individuals use positive emotions to bounce back from negative emotional experiences. *Journal of Personality and Social Psychology*, 86(2), 320–333. <a href="https://doi.org/10.1037/0022-3514.86.2.320">https://doi.org/10.1037/0022-3514.86.2.320</a>
- Zwarenstein, M., Goldman, J., & Reeves, S. (2009). Interprofessional collaboration: Effects of practice-based interventions on professional practice and healthcare outcomes. *Cochrane Database of Systematic Reviews, Issue 3*. https://doi.org/10.1002/14651858.CD000072.pub2
- Wei, H., Hardin, S. R., & Watson, J. J. I. j. o. n. s. (2021). A unitary caring science resilience-building model: Unifying the human caring theory and research-informed psychology and neuroscience evidence. 8(1), 130-135. <a href="https://doi.org/10.1016/j.ijnss.2020.11.003">https://doi.org/10.1016/j.ijnss.2020.11.003</a>
- Collins, S. (2005). Stress management interventions for nurses: A systematic review. *Journal of Nursing Research*, 10(3), 45–60.
- Lazarus, R. S., & Folkman, S. (1987). Stress, appraisal, and coping. Springer Publishing Company.

### **APPENDIX** (1):

### **Boucher of**

### Nurses Stress Self-Care Educational Program (NSSCEP)

# Session 04.

### **Teamwork / Physical** Wellness

### **Enhance team cohesion and** personal well-being.

- Recognize your team contribution (e.g., empathy, attention to detail).
- Build trust using active listening, empathy, or open communication.
  - Identify, Understand, Suggest, Decide, Act, Apply team problem-solving (6 steps: Follow Up).
- Set boundaries (e.g., no work emails after 7
- Develop a follow-up plan:
- Weekly self-assessment (e.g., stress rating)
  - Skill practice (e.g., deep breathing)
- Peer check-ins and progress logging Enhance communication:
- Active listening (e.g., nodding, eye contact).
  - Empathetic listening (e.g., reflect feelings) Positive non-verbal cues (e.g., open
- Strategic questions (e.g., open-ended).

## **How to Use This**

## **Brochure**

- Review skills weekly to track progress.
- Use reflection worksheets to note challenges and successes.
- Share insights with mentors/peers during check-ins.
  - loin the NSSCEP WhatsApp group for ongoing support.
- Revisit regularly to sustain self-care and resilience

# **Self-Care Logbook**

Baily Checklists: Mark skills used (e.g., Deep Frack progress with the logbook: Breathing) and note impact.

- Weekly Check-In: Rate stress/resilience 1–10); reflect on strategies.
  - Peer Support: Log WhatsApp/colleague nteractions.
- Final Reflection: Summarize progress after 1 Contact researcher via participant card. month. Submit logbook after 1 month.



## Benefits

- Reduced stress and burnout
- Stronger team cohesion and patient care Enhanced resilience and job satisfaction
  - Certificate upon completion

manager for session schedules. Your care for others starts with self-care. Take charge of your well-being! Coordinate with your nursing - Join Us





abusuqair@gmail.com AMMAN - JORDAN

### **Nurses' Stress Self-**Program (NSSGED Care Educationa Brochu &

manage occupational stress and nurses in Jordanian hospitals to A guide for paediatric oncolog prevent burnout.



# Why This Program?

- emotional challenges can lead to demanding. High workloads and Paediatric oncology nursing is burnout. This program helps nurses:
- Manage stress and burnout symptoms
- Build resilience with evidence-based tools
  - Strengthen teamwork and communication
- Protect personal time and advocate for improvements

# **Program Structure**

month booster and WhatsApp weeks, led by an expert, with a 1peer support. Sessions fit busy Four 2-hour sessions over 2 nospital schedules.

# Session 01.

## Self-Care for Nurses

## Learn to manage occupational stress and prevent burnout.

- burnout (Maslach, 2016), identifying sources like high workload or night Define stress (WHO, 2021) and
- mpact on health and performance. neadache, irritability) and their Recognize symptoms (e.g.,
  - Apply coping strategies:
- Emotion-focused (e.g., talking to Problem-focused (e.g., setting boundaries).
- Reflect on one stress symptom and coping strategy in worksheets. a colleague).

### Session 02. **Strengthening Inner** Resources

## Learn to manage occupational stress and prevent burnout.

- Practice stress management:
- Deep Breathing (4-7-8, 3 rounds)
- Progressive Muscle Relaxation (5
- Eisenhower Matrix for time 0
- 5-4-3-2-1 grounding technique. management.
- Write optimistic thoughts (e.g., "I Enhance resilience: handled it well")
  - Use problem-solving (Identify, Analyze, Plan, Act).
- Build support networks via peer 0
  - debriefing. Link tasks to values (e.g., 0
- compassion).
- Practice self-compassion (e.g., "I'm doing my best").
  - Reframe negative thoughts (e.g., "I'm failing" to "I'm learning") using CBT echniques.



## Session (

## **Reframing Stress Thoughts**

## Foster positive thinking and resilience to manage stress.

- catastrophizing) with positive self-talk. Counter negative thoughts (e.g.,
  - Use daily affirmations (e.g., "I am Apply positive scripts (e.g., "I can capable").
    - Seek positive influences (e.g., manage this")
- Practice gratitude via 3 Good Things ournal (3 times/week) supportive mentors)
  - Build resilience:
- Record small wins (e.g., "Comforted a patient").
  - Assess and shift negative self-talk. 0
    - Use Brief Resilience Scale to identify growth areas.



### **APPENDIX (2):**

### Daily Logbook of

### Nurses Stress Self-Care Educational Program (NSSCEP)

### NSSCEP Skills Checklist: Stress Management & Burnout Prevention

This brochure summarizes key skills from the Nurses Stress Self-Care Educational Program (NSSCEP) to help paediatric oncology nurses in Jordanian hospitals manage occupational stress and prevent burnout. Use it to confirm your application of these evidence-based techniques, practiced over three days across two weeks, with a one-month booster and peer support via WhatsApp. Refer to your reflection worksheets for detailed tracking.

| Participant Code/Hospital:(e.g., I-A-1) | Week:(Insert Week Number or Date) |
|---|---|
| Session 1: Self-Care Skills | Session 3: Positive Thinking |
| Recognize Stress/Burnout: Identify one symptom (e.g., eadache, irritability) and its impact. Identify Stressors: Name one workplace stressor (e.g., igh workload, night shifts). Apply Coping Strategies: Use one problem-focused (e.g., etting boundaries) or emotion-focused (e.g., talking to a bleague) strategy. Session 2: Resilience & Coping Stress Management Techniques: Deep Breathing (4-7-8, 3 rounds). Progressive Muscle Relaxation (5 min). Grounding (5-4-3-2-1 technique). Build Resilience: Write one optimistic thought (e.g., I handled it well). Use problem-solving (Identify, Analyze, Plan, Act). Connect with a colleague for support. Link a task to a value (e.g., compassion). Self-Compassion: Write/say a kind message (e.g., Im doing my best). Cognitive Restructuring: Reframe a negative thought (e.g., Im failing to Im learning). | <ul> <li>□ Positive Thinking:</li> <li>□ Counter one negative thought (e.g., catastrophizing).</li> <li>□ Use a daily affirmation (e.g., I am capable).</li> <li>□ Apply a positive script (e.g., I can manage this).</li> <li>□ Seek a positive influence (e.g., supportive mentor).</li> <li>□ Gratitude Practice: Write 3 Good Things daily, 3 times/week.</li> <li>□ Resilience Activities:</li> <li>□ Record a small win (e.g., Comforted a patient).</li> <li>□ Assess and shift negative self-talk.</li> <li>□ Use Brief Resilience Scale for growth areas.</li> <li>Session 4: Teamwork &amp; Well-Being</li> <li>□ Team Contribution: Recognize one strength (e.g., empathy).</li> <li>□ Trust &amp; Respect: Use one technique (e.g., active listening).</li> <li>□ Team Problem-Solving: Apply one step (e.g., identify a problem like delayed medication).</li> <li>□ Set Boundaries: Set one boundary (e.g., no emails after 7 PM).</li> <li>□ Follow-Up Plan: Log one action (e.g., stress rating).</li> </ul> |
| | <ul> <li>□ Communication Skills:</li> <li>□ Use active listening (e.g., nodding, eye contact).</li> <li>□ Apply empathetic listening (e.g., reflect feelings).</li> <li>□ Use positive non-verbal cues (e.g., open posture).</li> <li>□ Ask a strategic question (e.g., open-ended).</li> </ul> |
| Reflection | |
| <ul> <li>What worked well? Note a skill or moment that reduced st</li> </ul> | [171-11] |

• Next weeks plan: Choose one skill to focus on (e.g., gratitude). [Use worksheet]

### How to Use This Checklist?

- · Check off skills you've applied each week to confirm progress.
- Share reflections with a mentor/peer during weekly check-ins (Sessions 2, 4).
- Use communication skill checklists for interactions.
- · Revisit weekly to sustain self-care and prevent burnout.
- Contact your facilitator for support or join the NSSCEP WhatsApp group.

Your dedication in paediatric oncology nursing makes a difference. Prioritize your well-being to sustain compassionate care.

## General Safety Programme for Control Group Teaching Quid

22/8/2025

### **CONTROL GROUP PROGRAM**

### DAY ONE / 2 HOURS

| Session 1: Infection Prevention and Hand Hygiene | | | | | |
|---|---|---|---|---|---|
| Objective | | Content (Topics) | Materials/Aids | T | eaching strategy |
| Reinforce awareness and adherence to infection control and hand hygiene standards in pediatric oncology settings. | <ol> <li>3.</li> <li>4.</li> </ol> | WHO's Five Moments for Hand Hygiene Correct handwashing techniques (soap and alcohol-based rub) Use of gloves and personal protective equipment (PPE) Preventing infection in immunocompromised | Laptop and projector WHO guidelines Video Show Handout summarizing infection control procedures | 3. | Short lecture and Video demonstration Live hand hygiene practice Group discussion on local hospital practices Simulation exercise, debriefing discussion. |
| Session | 2: 1 | Hospital Safety and Emergen | cv Protocols | | |
| Objective | | ı Ü | Materials/Aids | T | eaching strategy |
| Improve nurse preparedness in responding to safety hazards and emergency situations. | | principles Emergency codes (e.g., Code Blue, Code Red) Evacuation routes and procedures Electrical, chemical, and radiation safety Safe patient handling and fall prevention | projector Safety code chart Scenario-based worksheet | <ol> <li>1.</li> <li>2.</li> <li>3.</li> </ol> | Interactive lecture<br>Quiz game on<br>safety codes<br>Facility map<br>discussion |

### **CONTROL GROUP PROGRAM**

### DAY TWO / 2 HOURS

| Session 3: Optimizing Workflow Documentation and Quality Control Medication Administration | | | | | |
|---|---|---|---|---|---|
| Objective | | Content (Topics) | Materials/Aids | T | eaching strategy |
| Enhance efficiency in daily nursing responsibilities through better documentation and medication practices in Jordanian settings, focusing on technical accuracy. | | Optimizing documentation: Best practices for electronic health records Strategies for efficient charting software use The Five Rights of medication administration Paediatric dosing principles and calculations Common causes of medication errors Reporting errors and near misses Safe storage and labelling. | Medication<br>error report<br>form (sample),<br>video show,<br>flip chart, case<br>scenarios for<br>prioritization<br>practice,<br>worksheet,<br>whiteboard or<br>flip chart,<br>projector. | <ol> <li>2.</li> <li>3.</li> </ol> | activity. Casebased simulation. Group debriefing. |
| Session 4: P | | essional Ethics in Paediatric | Oncology Nursi | ng | |
| Objective | | Content (Topics) | Materials/Aids | | eaching strategy |
| Refresh understanding of core ethical principles in clinical decision-making and care delivery. | <ol> <li>3.</li> </ol> | Confidentiality and patient rights Informed consent in paediatrics Boundaries in nurse—child—parent relationships Advocacy and best interest of the child Ethical dilemmas in paediatric oncology care | Laptop and projector ANA Code of Ethics summary Discussion prompts | | Short lecture Small group discussion of ethical cases Role-play (nurse- parent-child scenarios) Debriefing and summary |

### **Control Group Programme: Professional Skills Enhancement Programme**

### **Overview**

The Professional Skills Enhancement Programme is designed to refresh and strengthen essential technical skills for Jordanian paediatric oncology nurses, ensuring high-quality care delivery while serving as a placebo intervention. The programme consists of four 2-hour sessions over two days, delivered by a trained facilitator using a detailed script to maintain a neutral, didactic tone, with session fidelity monitored via recorded samples and a fidelity checklist to ensure no stress-related content is introduced. It is coordinated with nursing managers to align with shift schedules and avoid peak stress periods (e.g., holidays). Sessions are offered in flexible formats (in-person or recorded virtual access), with personalised WhatsApp reminders and verbal endorsements from nurse leaders to prevent dropout.

Participants receive printed handouts, a certificate of appreciation with specific skill endorsements (e.g., "Certified in Paediatric Oncology Safety") and potential continuing education credits (CECs), subject to hospital approval, to enhance perceived value. A peer support WhatsApp group facilitates skill sharing without discussing stress or emotions, and a 3-month booster session (1 hour, virtual or in-person) reinforces skills. The programme is culturally relevant, addressing Jordanian hospital realities (e.g., resource constraints, family dynamics), and matches the experimental group's contact time and engagement level.

### **Session 1: Infection Prevention and Hand Hygiene (1 Hours)**

- 1. Hospital-Acquired Infections (HAIs): Define HAIs (e.g., catheter-associated bloodstream infections, ventilator-associated pneumonia) and their impact in paediatric oncology, including increased morbidity and hospital costs. Highlight prevalence in developing countries like Jordan, where resource constraints exacerbate risks (Allegranzi et al., 2011). Discuss the roles of nurses in prevention.
- 2. WHO's Five Moments for Hand Hygiene: Explain the five critical moments: before touching a patient, before clean/aseptic procedures, after body fluid exposure risk, after touching a patient, and after touching patient surroundings. Provide examples from Jordanian hospitals (e.g., central line dressing changes) to illustrate application (World Health Organization, 2009).
- 3. **Correct Handwashing Techniques:** Demonstrate soap-and-water washing (20–40 seconds) and alcohol-based hand rub (15–20 seconds), covering all hand surfaces (palms, fingers, thumbs, wrists). Address common errors and barriers (e.g., limited water supply in some facilities).
- 4. **Use of Gloves and Personal Protective Equipment (PPE):** Detail protocols for selecting, donning, and doffing gloves, masks, gowns, and eye protection in oncology wards. Discuss safe disposal and reuse challenges in Jordanian settings. Include chemotherapy-specific PPE requirements.
- 5. **Preventing Infection in Immunocompromised Children:** Outline strategies like environmental cleaning, sterile technique for invasive procedures, and visitor restrictions. Emphasise nurse advocacy for infection control policies in resource-limited settings.
- 6. Hand Hygiene Simulation with UV Gel: Practical exercise using UV gel under blacklight to visualise missed areas, followed by group discussion on improving technique. Participants create a personal hand hygiene checklist for daily use.

7. **Case Study Analysis:** Review a Jordanian hospital case (e.g., HAI outbreak due to poor hand hygiene) to identify prevention strategies, reinforcing practical application.

### **Notes for Facilitators**

- Maintain a neutral tone, framing content as technical skill enhancement (e.g., "improving patient safety" rather than "reducing infection-related stress").
- Use Jordanian hospital examples (e.g., King Hussein Cancer Center protocols) to ensure relevance.
- Encourage participation in simulations but avoid probing personal experiences or emotions.
- Monitor group dynamics to ensure quieter participants engage during case study discussions; assign roles (e.g., note-taker) if needed.
- Reinforce the value of CECs and certificates to motivate completion.

### **Discussion Points**

- What are common barriers to hand hygiene in your Jordanian hospital (e.g., time constraints,
   PPE shortages)? How can nurses address these within existing resources?
- How do visitor policies in Jordanian oncology wards impact infection control? Share practical enforcement strategies.
- Based on the case study, what specific actions could nurses take to prevent similar HAIs in your workplace?

### **Session 2: Hospital Safety and Emergency Protocols (1 Hours)**

- 1. Fire Safety (PASS and RACE Principles): Explain PASS (Pull, Aim, Squeeze, Sweep) for fire extinguisher use and RACE (Rescue, Alarm, Confine, Extinguish/Evacuate) for fire response. Highlight fire risks in oncology wards (e.g., oxygen tanks, chemotherapy storage) and Jordanian hospital compliance requirements (Joint Commission International, 2020).
- **2. Emergency Codes:** Detail hospital-specific codes (e.g., Code Blue for cardiac arrest, Code Red for fire, Code Pink for infant abduction). Clarify nurse roles, communication protocols, and documentation during emergencies in Jordanian settings.
- **3. Evacuation Routes and Procedures:** Review hospital evacuation plans, prioritising immunocompromised patients and using safe routes. Discuss challenges such as crowded corridors or limited lifts in Jordanian facilities.
- **4. Electrical, Chemical, and Radiation Safety:** Outline protocols for managing electrical faults, chemical spills (e.g., chemotherapy drugs), and radiation exposure risks. Emphasise proper labelling, storage, and spill kits in oncology units.
- **5. Safe Patient Handling and Fall Prevention:** Teach techniques for transferring paediatric patients and preventing falls (e.g., bed rails, non-slip flooring). Address risks for weak or sedated children in oncology care.
- **6. Mock Emergency Drill Using Jordanian Facility Maps:** Group activity to simulate a Code Red response, using hospital-specific maps to plan evacuation routes, assign roles, and identify bottlenecks.
- **7. Safety Audit Checklist Development:** Participants create a ward-specific safety checklist (e.g., checking fire exits, equipment storage) for daily use.

### **Notes for Facilitators**

- Focus on procedural knowledge (e.g., "follow RACE steps") rather than emotional preparedness.
- Use hospital-specific maps to ground activities in local context, enhancing relevance.
- Ensure drills remain technical; avoid discussing fear or stress during emergencies.
- Encourage equal participation in group activities by assigning roles (e.g., leader, scribe).
- Highlight practical benefits of checklists for daily ward routines to motivate adoption.

### **Discussion Points**

- What safety hazards are most common in your Jordanian oncology ward (e.g., cluttered corridors, faulty equipment)? How can nurses address these?
- How do emergency codes function in your hospital? Share examples of effective code responses.
- Based on the mock drill, what improvements could be made to your ward's evacuation plan?

### Session 3: Optimising Workflow Documentation and Medication Administration (1 Hours)

- 1. Optimising Electronic Health Records (EHRs): Review best practices for accurate, timely EHR entries using structured templates and mandatory fields. Discuss Jordanian systems like Hakeem, common errors (e.g., incomplete fields), and their impact on care continuity (Kalra, 2011).
- **2. Actionable Shift Reports:** Teach SBAR (Situation, Background, Assessment, Recommendation) for concise handovers. Provide examples tailored to paediatric oncology (e.g., reporting chemotherapy side effects).
- **3. Efficient Charting Software Use:** Share tips for navigating EHR interfaces, using shortcuts, and resolving technical issues (e.g., system downtime). Address challenges in Jordanian hospitals, such as slow connectivity.
- **4. Five Rights of Medication Administration:** Ensure the right patient, drug, dose, route, and time through verification (e.g., barcode scanning, double-checking). Discuss oncology-specific risks (e.g., chemotherapy errors).
- **5.** Paediatric Dosing Principles and Calculations: Review weight-based dosing for chemotherapy and supportive drugs, using Jordanian formularies. Practice calculations with real-world examples (Cohen, 2015).
- **6.** Common Causes of Medication Errors: Identify risks (e.g., look-alike drugs, illegible orders) and prevention strategies (e.g., standardised protocols, clear labelling).
- **7. Reporting Errors and Near Misses:** Outline non-punitive reporting protocols in Jordanian hospitals, encouraging transparency to improve safety.

- **8. Safe Storage and Labelling:** Discuss storage of high-risk medications (e.g., chemotherapy agents) and tamper-evident labelling to prevent misuse.
- **9. Group Prioritisation Simulation with Jordanian Sample Shift Schedules:** Activity to prioritise tasks (e.g., charting vs. medication rounds) using realistic Jordanian shift scenarios, followed by debriefing.
- **10. Documentation Workflow Mapping:** Participants map their current documentation process, identify inefficiencies, and propose improvements for their ward.

### **Notes for Facilitators**

- Frame activities as procedural optimisation (e.g., "streamline charting" not "reduce workload stress").
- Use familiar Jordanian systems (e.g., Hakeem) to ensure applicability.
- Provide clear instructions for calculations to avoid confusion, offering examples first.
- Ensure simulations focus on task prioritisation, not emotional responses to workload.
- Encourage participants to share workflow tips but redirect if discussions veer into stress complaints.

### **Discussion Points**

- How does your hospital's EHR system (e.g., Hakeem) support or hinder efficient documentation? Share practical tips for improvement.
- What strategies ensure the Five Rights during busy shifts in Jordanian oncology wards?
- Based on the prioritisation simulation, how can your team better organise tasks during peak hours?

### Session 4: Professional Ethics in Paediatric Oncology Nursing (1 Hours)

- Confidentiality and Patient Rights: Review Jordanian legal and hospital policies on privacy, including handling sensitive data (e.g., cancer diagnoses) and communicating with families. Discuss cultural expectations around family involvement (Fry & Johnstone, 2008).
- 2. **Informed Consent in Paediatrics:** Outline the consent process for parents/guardians, including explaining risks and benefits in culturally sensitive ways. Address assent from older children and legal considerations in Jordan.
- 3. **Boundaries in Nurse-Child-Parent Relationships:** Provide guidelines for maintaining professional boundaries while showing compassion, avoiding over-involvement or favouritism. Discuss cultural norms in Jordanian family dynamics.
- 4. **Advocacy for the Child's Best Interest:** Explore nurse roles in advocating for patient needs (e.g., pain management, psychosocial support) within teams and family contexts. Highlight advocacy within resource constraints.
- 5. **Ethical Dilemmas in Jordanian Paediatric Oncology:** Discuss common dilemmas (e.g., parental refusal of treatment due to cost, withholding care due to resource shortages) and apply decision-making frameworks (e.g., autonomy, beneficence).
- 6. **Role-Play for Ethical Scenarios with Jordanian Families:** Simulate ethical challenges (e.g., discussing treatment refusal, managing family conflicts), using culturally relevant scenarios with props (e.g., mock charts).
- 7. **Ethical Decision-Making Framework Development:** Participants create a personal decision-making guide based on ethical principles, tailored to their ward's challenges.

### **Notes for Facilitators**

- Keep discussions focused on ethical principles and procedures, not emotional responses to dilemmas.
- Use culturally sensitive scenarios (e.g., family-driven decision-making in Jordan) to enhance relevance.
- Ensure role-plays remain professional; redirect if participants discuss personal distress.
- Assign roles in group activities to ensure inclusivity, especially for less vocal participants.
- Emphasise the practical utility of decision-making guides for daily practice.

### **Discussion Points**

- How do Jordanian cultural norms (e.g., family involvement) shape informed consent processes in your ward?
- What ethical dilemmas have you observed in Jordanian oncology care? How were they resolved?
- Based on the role-play, what strategies can nurses use to navigate family conflicts while maintaining professionalism?

### References

Allegranzi, B., Nejad, S. B., Combescure, C., Graafmans, W., Attar, H., Donaldson, L., & Pittet, D. (2011). Burden of endemic health-care-associated infection in developing countries: Systematic review and meta-analysis. *The Lancet*, 377(9761), 228–241. https://doi.org/10.1016/S0140-6736(10)61458-4

Cohen, M. R. (2015). *Medication errors* (2nd ed.). American Pharmacists Association. ISBN: 978-1582120928

Fry, S. T., & Johnstone, M.-J. (2008). *Ethics in nursing practice: A guide to ethical decision making* (3rd ed.). Wiley-Blackwell. ISBN: 978-1405160520

Institute for Safe Medication Practices. (2020). *ISMP list of high-alert medications in acute care settings*. <a href="https://www.ismp.org/recommendations/high-alert-medications-acute-list">https://www.ismp.org/recommendations/high-alert-medications-acute-list</a>

Joint Commission International. (2020). *International patient safety goals*. https://www.jointcommissioninternational.org/standards/international-patient-safety-goals/

Kalra, J. (2011). *Medical errors and patient safety: Strategies to reduce and disclose medical errors and improve patient safety*. De Gruyter. ISBN: 978-3110249491

Situation, Background, Assessment, Recommendation (SBAR) Toolkit. (2018). Institute for Healthcare Improvement. <a href="http://www.ihi.org/resources/Pages/Tools/SBARToolkit.aspx">http://www.ihi.org/resources/Pages/Tools/SBARToolkit.aspx</a>

World Health Organization. (2009). *WHO guidelines on hand hygiene in health care*. <a href="https://www.who.int/publications/i/item/9789241597906">https://www.who.int/publications/i/item/9789241597906</a>